CLINICAL TRIAL: NCT03232450
Title: PFOCUS Pilot Trial- A Prospective Pilot Trial for PFO ClosUre at the Time of endovaScular Cardiac Electronic Device Implantation
Brief Title: Patent Foramen Ovale (PFO) Closure at the Time of Endovascular Cardiac Electronic Device Implantation
Acronym: PFOCUS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding or enrollment
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Samuel J. Asirvatham, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-005348
Record Dates: First submitted 2017-07-20; First posted 2017-07-28 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Foramen Ovale, Patent
MeSH Terms: conditions — Foramen Ovale, Patent | interventions — Aspirin; Device Lead Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- PFO Closure (Active Comparator): Subjects randomized to this arm will receive 81 mg enteric coated aspirin, a Cardiovascular Implantable Device (CIED), Gore Cardioform Septal Occluder.
  Interventions: Drug: Aspirin; Device: Cardiovascular Implantable Device (CIED); Device: Gore Cardioform Septal Occluder
- Control (Other): Subjects randomized to this arm will receive 81 mg enteric coated aspirin, a Cardiovascular Implantable Device (CIED)
  Interventions: Drug: Aspirin; Device: Cardiovascular Implantable Device (CIED)

INTERVENTIONS:
Drug: Aspirin — Subjects will receive 81 mg enteric coated aspirin
  Other Names: Acetylsalicylic acid (ASA)
Device: Cardiovascular Implantable Device (CIED) — All subjects will receive either a pacemaker, implantable cardioverter-defibrillator (ICD), or cardiac resynchronization therapy (CRT).
Device: Gore Cardioform Septal Occluder — The Gore Cardioform Septal Occluder closes the patent foramen ovale (PFO).
  Arms: PFO Closure

SUMMARY:
Participants enrolled in this study will have been diagnosed with patent foramen ovale (PFO) and have been scheduled to have a cardiovascular implantable electronic device (CIED) such as a pacemaker, implantable cardioverter-defibrillator (ICD), or cardiac resynchronization therapy (CRT) device implanted. A PFO is a condition when there is a hole in the septum (the wall separating the right and left sides) of the heart.

The purpose of this study is to determine whether closing the PFO with the GORE® Cardioform Septal Occluder in people with an endocardial device leads reduces the risk of recurrent stroke or imaging-confirmed transient ischemic attack (TIA) compared to not closing the PFO.

ELIGIBILITY:
Inclusion Criteria:

* A clinical indication for a transvenous pacemaker or defibrillator implantation,
* Must have a documented PFO determined from Transthoracic Echocardiogram (TTE) echocardiographic agitated saline contrast study that is determined to be feasible for transcatheter closure.
* The GORE® CARDIOFORM Septal Occluder should only be used in subjects whose vasculature is adequate to accommodate a 10 Fr delivery sheath (or 12 Fr delivery sheath when a guidewire is used).
* All subjects must be able to undergo standardized neurocognitive testing, and dementia/mental status examination screening.

Exclusion Criteria:

* Subjects with a survival expectancy of less than one year.
* Subjects with an atrial septal defect or shunt that clinically requires closure for hemodynamic or other purposes.
* Absence of a clinical indication for a transvenous CIED system.
* Subjects with any clinical indication mandating anticoagulation.
* Subjects with previously placed CIED devices will be excluded.
* Unable to take anti-platelet medications such as aspirin or clopidogrel (Plavix).
* With anatomy where the GORE® CARDIOFORM Septal Occluder size or position would interfere with other intracardiac or intravascular structures, such as cardiac valves or pulmonary veins.
* With active endocarditis, or other infections producing bacteremia, or with known sepsis within one month of planned implantation, or any other infection that cannot be treated successfully prior to device placement.
* With known intracardiac thrombi.
* Known pregnancy at the time of automated implantable cardioverter-defibrillator (AICD) implant

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of Embolic Brain Lesions Detected on MRI >3 mm | 1 year post implantation
  The mean number of embolic brain lesions will be calculated at approximately 1 year.

SECONDARY OUTCOMES:
Number of Subjects Who Die | 1 year post implantation
  The mean number of deaths will be calculated at approximately 1 year.
Number of Subjects Who Experience a Stroke | 1 year post implantation
  Stroke is defined as an acute episode of focal or global neurological dysfunction caused by brain, spinal cord, or retinal vascular injury as a result of hemorrhage or infarction.
Number of Subjects who Experience a Transient Ischemic Attack (TIA) | 1 year post implantation
  Transient ischemic attack (TIA) is defined as a transient episode of focal neurological dysfunction caused by brain, spinal cord, or retinal ischemia, without acute infarction.
Change in Executive Function as Measured by Trail Making Test B | baseline, 1 year post implantation
  Trail Making Test B consists of 25 circles including both numbers (1-13) and letters (A-L). The subject draws lines to connect the circles in an ascending pattern, but with the added task of alternating between the numbers and letters. The subject is timed as they draw the trail. Results are reported as the number of seconds required to complete the task; therefore, higher scores reveal greater impairment. The average score is 75 seconds; > 273 seconds is considered deficient.
  Trail Making Test B consists of 25 circles including both numbers (1 - 13) and letters (A - L). The subject draws lines to connect the circles in an ascending pattern, but with the added task of alternating between the numbers and letters. The subject is timed as they draw the trail. Results are reported as the number of seconds required to complete the task; therefore, higher scores reveal greater impairment. The average score is 75 seconds; > 273 seconds is considered deficient.
Change in Language as Measured by Letter and Category Fluency Test | baseline, 1 year post implantation
  The examiner gives the subject a category and ask them to name all the different examples that they can think of from that category in one minute. Examples of categories are animals, fruit, birds, breeds of dog, tools, etc. Subjects are also asked to provide examples that start with a given letter. To score, the examiner counts the number of unique responses for a category or letter for one minute; categories can be averaged together. The higher the score the better the language fluency, the lower the score, the worse the language fluency.
Change in Psychomotor Speed as Measured by Trail Making A Test | baseline, 1 year post implantation
  Trail Making Test A consists of 25 numbered circles distributed over a sheet of paper. The patient should draw lines to connect the numbers in ascending order. The patient is timed as they draw the trail. Results are reported as the number of seconds required to complete the task; therefore, higher scores reveal greater impairment. The average score is 29 seconds; > 78 seconds is considered deficient.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel J Asirvatham, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials